CLINICAL TRIAL: NCT07254728
Title: A Phase I, Multicenter, Randomized, Double-blind, Placebo-controlled Single Dose, Dose-ranging Study to Evaluate the Safety, Tolerability, and Immunogenicity of Orally Administered Bivalent GI.1/GII.4 Norovirus Vaccine in Healthy Lactating Females ≥ 18 Years Old and Their Breast-feeding Infants
Brief Title: A Study to Evaluate Vaxart's Oral Bivalent GI.1/GII.4 Norovirus Vaccine in Healthy Lactating Females and Their Nursing Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VXA-NVV-108
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Norovirus Infections
Keywords: Healthy participants; VXA-G1.1-NN; VXA-G2.4-NS
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bivalent GII.4/GI.1 Medium Dose Vaccine (Experimental): Participants will receive a medium dose of bivalent VXA-G1.1-NN and VXA-GII.4-NS as an oral tablet on Day 1.
  Interventions: Biological: VXA-G1.1-NN; Biological: VXA-G2.4-NS
- Bivalent GII.4/GI.1 High Dose Vaccine (Experimental): Participants will receive a high dose of bivalent VXA-G1.1-NN and VXA-GII.4-NS as an oral tablet on Day 1.
  Interventions: Biological: VXA-G1.1-NN; Biological: VXA-G2.4-NS
- Placebo (Placebo Comparator): Participants will receive matching placebo orally on Day 1.
  Interventions: Biological: Placebo Tablets

INTERVENTIONS:
Biological: VXA-G1.1-NN — Oral tablets.
  Other Names: GI.1
  Arms: Bivalent GII.4/GI.1 High Dose Vaccine; Bivalent GII.4/GI.1 Medium Dose Vaccine
Biological: VXA-G2.4-NS — Oral tablets.
  Other Names: GII.4
  Arms: Bivalent GII.4/GI.1 High Dose Vaccine; Bivalent GII.4/GI.1 Medium Dose Vaccine
Biological: Placebo Tablets — Oral tablets.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of an oral bivalent GI.1/GII.4 norovirus vaccine administration in healthy lactating female participants and to assess the short-term immunogenicity of oral bivalent GI.1/GII.4 norovirus vaccine administration in healthy lactating female participants and its association with the immunogenicity response in breastmilk.

ELIGIBILITY:
Inclusion Criteria:

1. Lactating females aged ≥ 18 years at the time of enrolment and their breastfed infants aged >30 days to 11 months of age at the time of the participants' study drug administration.
2. In stable and good general health, without significant medical illness, based on medical history, physical examination (including vital signs), and clinical judgment of the investigator.
3. Lactating females willing and able to provide informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
4. Lactating females who are willing to provide consent for their breastfed infant.
5. Negative pregnancy tests at screening and prior to dose on Day 1.
6. Available for all planned visits and tele-health appointments, and ability to comply with all study-related evaluations (including but not limited to having the ability and willingness to swallow multiple small enteric-coated tablets per study dose, express/pump breastmilk, and collect infant stool samples).
7. Plan to continue breastfeeding as the main source of the infant's nutrition for at least 1 month (longer is preferred with goal of 6 months post dose if possible) from the time of study drug administration. Exclusive breastfeeding is acceptable but not necessary.
8. The nursing infant is the product of a singleton pregnancy AND does not have any of the following:

   1. Any abnormality that may interfere with breastfeeding or milk absorption
   2. Active infection (may be included if the infection resolves and the participant is re-assessed during the screening period)
   3. Infant has any other medical condition or abnormality that, in the opinion of the investigator, could compromise the infant's appropriate inclusion in this study including interference with the interpretation of study results (such as malabsorption)
   4. One or more documented brief resolved unexplained events (BRUEs)
   5. Extreme prematurity (infants who were born at less than 28 weeks gestation)
   6. 30 days of age or less at the participant's study drug administration OR greater than 11 months of age at the participant's study drug administration
   7. Prior hospitalization that is not exclusively for hyperbilirubinemia requiring phototherapy
   8. Any genetic/metabolic disease
   9. Any chronic illness requiring long term medication
9. Participants must be willing to use a highly effective form of contraception for 30 days prior to vaccination and until 60 days after the vaccination. Acceptable forms are oral, implantable, intrauterine, transdermal, intravaginal, injectable, double barrier or abstinence (participants using diaphragms must also use condom). The form of contraception must be approved by the investigator.

Exclusion Criteria:

1. Presence of a fever ≥ 38.0°C measured orally at baseline, on Day 1 prior to vaccination. (Assessment may be repeated once during screening period).
2. Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam). (Assessment may be repeated once during screening period).
3. Participants who have received antipyretic/analgesic medications within 24 hours prior to the intended vaccine administration.
4. Positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) tests at the screening visit.
5. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin.
6. History of serious reactions to vaccination such as anaphylaxis, respiratory problems, hives, or abdominal pain.
7. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including the institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline.
8. History of significant pregnancy-related complications during this pregnancy, including but not limited to pre-eclampsia, eclampsia, or gestational diabetes unless a full resolution is documented.
9. Cancer, or treatment for cancer, within the past 3 years (excluding fully treated and resolved basal cell carcinoma or squamous cell carcinoma).
10. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus type 1 or 2.
11. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine. Such conditions may include but are not limited to:

    a. Any history of:

    i. Malignancy

    ii. Malabsorption

    iii. Pancreatobiliary disorders

    iv. Inflammatory bowel disease

    v. Irritable bowel disease

    vi. Hiatal hernia

    vii. Surgical resection

    b. History of diagnosis or treatment in past 5 years of:

    i. Esophageal or gastric motility disorder

    ii. Gastroesophageal reflux disease (GERD) - Will allow for participants with a history of pregnancy-related GERD if fully resolved for >3 months and no other history of GERD diagnosis

    iii. Peptic ulcer

    iv. Cholecystectomy
12. Any condition that resulted in the absence or removal of the spleen.
13. History of any form of angioedema.
14. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic.
15. History of GI bleeding including hematochezia (blood in stool) or melena (black stool).
16. Any significant hospitalization within the last year which in the opinion of the investigator or sponsor could interfere with study participation.
17. Any of the following history or conditions that may lead to a higher risk of clotting events and/or thrombocytopenia:

    1. Family or personal history of bleeding or thrombosis
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments
    3. History of autoimmune or inflammatory disease
    4. Presence of any of the following conditions known to increase the risk of thrombosis within 6 months prior to screening:

    i. Recent surgery other than fully healed cesarean delivery or excision/ biopsy of cutaneous lesions

    ii. Immobility (confined to bed or wheelchair for 3 or more successive days)

    iii. Head trauma with loss of consciousness or documented brain injury

    iv. Receipt of anticoagulants for prophylaxis of thrombosis

    v. Recent clinically significant infection including hospitalization for COVID-19 related illness
18. Any other condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of a participant taking in the study, would render the participant unable to comply with the protocol, or would interfere with the evaluation of the study endpoints.
19. Receipt of a licensed vaccine (including any COVID-19 vaccines under Emergency Use Authorization) within 14 days prior to study drug dose or planned administration during the study active period.
20. Use of antibiotics, proton pump inhibitors, H2 blockers, or antacids within 7 days prior to study drug administration or planned use during the active study period.
21. Use of medications known to affect the immune function (including but not limited to systemic corticosteroids, leukotriene modifiers, and Janus kinase [JAK] inhibitors) within 2 weeks before study drug administration or planned use during the active study period.
22. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study drug administration or planned use during the active study period.
23. Donation or receipt of blood or blood products within 30 days prior to study drug administration or planned donation during the active study period.
24. Participating in any clinical trial with another investigational product within 30 days prior to the first trial visit or intend to participate in another clinical trial at any time during the conduct of this trial.
25. Are first-degree relatives of individuals involved in trial conduct.
26. Positive urine drug screen for drugs of abuse at screening.
27. Positive alcohol test at screening or baseline.
28. History of drug, alcohol, or chemical abuse within 1 year of screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Solicited Symptoms of Reactogenicity for 8 Days Post Dose | 1 week post study dose (8 days)
Number of Participants With Unsolicited Treatment-emergent Adverse Events (TEAEs) | 4 weeks post dose (29 days)
  Number of Participants With Unsolicited TEAEs includes participants with serious AEs (SAEs), adverse events of special interest (AESIs) and new onset of chronic illness (NOCIs).
Geometric Mean Concentration (GMC) at Day 1 of Serum Viral Protein 1 (VP1) Specific (GI.1 and GII.4) Immunoglobulin A (IgA) | Day 1
GMC at Day 8 of Serum VP1 Specific (GI.1 and GII.4) IgA | Day 8
GMC at Day 29 of Serum VP1 Specific (GI.1 and GII.4) IgA | Day 29
Geometric Mean Fold Rise (GMFR) From Day 1 to Day 8 of Serum VP1 Specific (GI.1 and GII.4) IgA | From Day 1 to Day 8
GMFR From Day 1 to Day 29 of Serum VP1 Specific (GI.1 and GII.4) IgA | From Day 1 to Day 29
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgA (GI.1 and GII.4) at Day 1 | Day 1
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgA (GI.1 and GII.4) at Day 8 | Day 8
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgA (GI.1 and GII.4) at Day 29 | Day 29
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgA (GI.1 and GII.4) at Day 60 | Day 60
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgA (GI.1 and GII.4) at Day 180 | Day 180
GMC at Day 1 of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 1
GMC at Day 8 of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 8
GMC at Day 29 of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 29
GMFR From Day 1 to Day 8 of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 1 to Day 8
GMFR From Day 1 to Day 29 of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 1 to Day 29
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater GMC Rise or Greater in Breastmilk VP1 Specific IgA (GI.1 and GII.4) at Day 1 | Day 1
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater GMC Rise or Greater in Breastmilk VP1 Specific IgA (GI.1 and GII.4) at Day 8 | Day 8
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater GMC Rise or Greater in Breastmilk VP1 Specific IgA (GI.1 and GII.4) at Day 29 | Day 29
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater GMC Rise or Greater in Breastmilk VP1 Specific IgA (GI.1 and GII.4) at Day 60 | Day 60
Number of Participants Who Achieve a 2-fold, 3-fold and 4-fold GMC Rise or Greater in Breastmilk VP1 Specific IgA (GI.1 and GII.4) at Day 180 | Day 180

SECONDARY OUTCOMES:
Number of Participants With SAEs, AESIs and NOCIs Through 12 months Post Dose | Up to 12 months
GMC of Serum VP1 Specific (GI.1 and GII.4) IgA | Day 180
GMFR of Serum VP1 Specific (GI.1 and GII.4) IgA | From Day 1 to Day 180
GMC of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | Day 60 and Day 180
GMFR of Breastmilk VP1 Specific (GI.1 and GII.4) IgA | From Day 1 to Day 180
GMC of Serum VP1 Specific (GI.1 and GII.4) IgG | Days 1, 8, 29 and 180
GMFR of Serum VP1 Specific (GI.1 and GII.4) IgG | From Day 1 to Day 180
Number of Participants With 2-fold, 3-fold and 4-fold GMC Rise or Greater in Serum VP1 Specific IgG (GI.1 and GII.4) | Days 1, 8, 29, and 180
Geometric Mean Titer (GMT) of Serum Blocking Titers 50 (BT50) (GI.1 and GII.4) | Days 1, 8, 29, and 180
GMFR of Serum BT50 (GI.1 and GII.4) | From Day 1 to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Vaxart, Inc.
Locations (5):
- South Africa (5):
  - WITS RHI Research Centre, Hillbrow
  - Progress Clinical Research Unit, Honeydew
  - Newtown Clinical Research Centre, Johannesburg
  - Trident Clinical, Kimberley
  - FCRN Clinical Trials Centre (Pty) Ltd, Vereeniging

IPD SHARING:
Plan to Share IPD: No